CLINICAL TRIAL: NCT03104920
Title: ERAS (Early Recovery After Surgery) Program Improve the Recovery of the Patient Undergoing Curative Hepatectomy: a Prospective Multicenter Cohort Trial
Brief Title: ERAS Program Improves Recovery of HCC Patient Undergoing Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: feng xiaobin (Other)
Responsible Party: Sponsor-Investigator, feng xiaobin, Associate Proffesor, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWHB016
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: HCC
Keywords: ERAS; Time to ready for discharge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS program (Experimental): We give an ERAS pathway, which comprises of optimized management of diet, mobilization, analgesia and GI function recovery for patients with HCC.
  Interventions: Procedure: ERAS Program
- Traditional treatment (Active Comparator): We give routine clinic practices for the treatment of HCC.
  Interventions: Procedure: Traditional treatment

INTERVENTIONS:
Procedure: ERAS Program — An ERAS pathway comprises of optimized management of diet, mobilization, multimodal perioperative analgesia and GI function recovery modalities.
  Arms: ERAS program
Procedure: Traditional treatment — A traditional perioperative management for HCC.
  Arms: Traditional treatment

SUMMARY:
The worldwide introduction of multimodal enhanced recovery programs has also changed perioperative care in patients who undergo liver resection. This study will be performed to assess a comprehensive care package for patients with hepatocellular carcinoma (HCC) undergoing hepatectomy with the aim of minimal physiological disturbance in the peri-operative period. Peri-operative opioid-sparing analgesia with few gastrointestinal (GI) effects and reduced requirement for intravenous fluid therapy, early ambulation and promoted GI function recovery were centered to this plan.

DETAILED DESCRIPTION:
The first ERAS program was introduced by Kehlet in the 1990's. ERAS programs were initially implemented in colorectal surgery and have found their way into general clinical practice, including orthopedic, vascular, and thoracic surgery. In the field of liver surgery, cohort studies have been conducted and randomized trials have confirmed the feasibility and safety of enhanced recovery programs in resectional liver surgery.

Randomized studies have suggested that ERAS optimization may contribute in decreasing stay in hospital after surgery. We hypothesized that opioid-sparing preemptive and post-operative multimodal analgesia plus other ERAS items would effectively accelerate patient recovery, who receiving hepatectomy. We focus on some fundamental variables that impact normal physiology and enhanced-recovery after surgery: fasting, opioid-sparing, exception of an abdominal drain, and GI function rehabilitation. We draw attention to the fact that time to recovery is a far more important and better outcome measure than time to discharge from the hospital.

GI function protection and restore was of importance as the respect of ERAS. Traditionally, perioperative fasting is consisted of being nil by mouth from midnight before surgery and fasting postoperatively until recovery of bowel function. Those empirical practices persist despite emerging evidence revealing that excessive fasting results in negative outcomes and delayed recovery. Strong and assistant evidence exists for minimization of perioperative fasting for 2-hour preoperative fast after clear fluids and for early oral food and fluids intake postoperatively. Also, current study should be applying anti-ileus prophylaxis and abolition of bowel preparation.

Optimizing pain control was regarding as one of the ultimate goal of ERAS program: pain and risk free surgery. Surgical incisions evoke nociceptors by inducing local inflammatory response. The consequence hyperalgesia has been considered to be target of well pain controlling. Here, the multimodal opioid-sparing approaches have been emphasized. A regimen composed by TAP, local anesthesia, PCA, and systematic anti-inflammatory would be performed in order to reduce surgical stress responses.

Several studies have reported that mobilization within 24h of colon surgery was an independent predictor of shorter rehabilitation period. In current study, early postoperative enforced mobilization with specific target will be implemented.

The purpose of this study is twofold. On the one hand examine the scientific evidence that exists today on the most important elements of an ERAS program and present preliminary results of the implementation of a program ERAS in West China.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent;
* Elective partial hepatectomy for HCC;
* No major concomitant surgical procedures such as bowl or bile duct resection;
* Tumors restricted in hepatic segment: II, III, IVb, VI and VII;
* Child-Pugh Class A/B liver function status；
* ECGO scores = 0

Exclusion Criteria:

* Tumor thrombi in portal vein;
* Tumor size >10cm;
* History of uncontrolled ascites, hepatic encephalopathy, and varices bleeding;
* ICG>14%;
* Concurrent with other malignant disease;
* Multiple organ dysfunctions;
* Viral infectious disease besides HBV and HCV;
* Diabetes Mellitus;
* Ruptured hepatocellular carcinoma;
* History of treatment such as TACE, RFI, PEI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
TRD (time to ready for discharge) | 1 month after surgery
  time to ready for discharge

SECONDARY OUTCOMES:
Readmission within 30 days of discharge | 30 days after surgery
  Readmission within 30 days of discharge
Complications rate | 3 months after surgery
  Complications rate
Postoperative LOS (length of hospital stay) | 30 days after surgery
  Postoperative length of hospital stay
Liver function recovery | 30 days after surgery
  Liver function recovery
Surgery Stress （CRP） | 15 days after surgery
  Surgery Stress indicated by c-reactive protein
Pain assessment（VAS，per day） | 3 months after surgery
  Pain assessment
Total cost | 3 months after surgery
  Total cost
Validated EQ-5D（EuroQol Group quantitum form） | 3 months after surgery
  Validated EQ-5D
First time of normal diet and stool passage | 7 days after surgery
  First time of normal diet and stool passage

CONTACTS AND LOCATIONS:
Overall Officials: Kuansheng Ma, Doctor, Study Director — Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No